CLINICAL TRIAL: NCT05489068
Title: Adapting Intake Procedures to Improve Treatment Delivery in Addiction Treatment
Brief Title: Motivational Interviewing at Intake vs Intake as Usual on Client Engagement in Addiction Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: A22-0014; K23DA052646 (NIH)
Record Dates: First submitted 2022-07-26; First posted 2022-08-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Substance-Related Disorders; Treatment Adherence
MeSH Terms: conditions — Substance-Related Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Effectiveness-Implementation Hybrid Type 1 Design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing at Intake (MII) (Experimental): Clients allocated to the MII condition will receive a 90-minute pure Motivational Interviewing (MI) session.
  Interventions: Behavioral: Motivational Interviewing at Intake (MII)
- Intake as Usual (IAU) (Active Comparator): Clients allocated to the IAU condition will receive the 90-minute standard assessment that is delivered to all clients entering intensive outpatient program (IOP)/outpatient program (OP).
  Interventions: Behavioral: Intake as Usual (IAU)

INTERVENTIONS:
Behavioral: Motivational Interviewing at Intake (MII) — The MII will involve a goal-oriented and collaborative conversation about why the client wants treatment now, and how treatment might fit with his/her most important values. The provider will use open questions, reflective listening and autonomy support in a flexible, non-authoritative manner. Rather than asking specific questions in different life domains, the provider will explore with the client their desires, abilities, reasons, and needs for treatment, how treatment fits with their values, and what successful treatment looks like to them. The client's language about change will be strategically reinforced to increase its frequency and strength across the session.
  Arms: Motivational Interviewing at Intake (MII)
Behavioral: Intake as Usual (IAU) — In line with the American Society of Addiction Medicine (ASAM) guidelines, the IAU condition involves a semi-structured interview of the client's psychosocial history and clients answer a series of questions in the following domains: support system, living situation, educational, occupational, family, and medical history.
  Arms: Intake as Usual (IAU)

SUMMARY:
This K23 study is an effectiveness-implementation hybrid type I design to determine the effectiveness of Motivational Interviewing at Intake (MII), relative to intake-as-usual on client engagement and mechanisms of engagement among adults seeking outpatient addiction treatment. We also will obtain personnel feedback on the feasibility of implementing MII into standard practice by having personnel from the addiction treatment study sites complete implementation climate measures before Motivational Interviewing (MI) training and post-clinical trial, as well as an individual interview on implementation feasibility post-trial.

ELIGIBILITY:
Inclusion Criteria (client participants):

* English-speaking adults seeking treatment for alcohol or other drug use at one of two outpatient addiction treatment programs
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures
* Physically withdrawn from alcohol or other drugs

Inclusion Criteria (personnel participants):

* English-speaking adults currently employed at one of the two outpatient addiction treatment programs
* Provision of electronic informed consent

Exclusion Criteria (client participants):

* Experiencing severe withdrawal symptoms
* Actively psychotic, manic, and/or suicidal

Exclusion Criteria (personnel participants):

* current position: facility owner or clinical director

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who attended the first outpatient treatment program session based on electronic medical record review | up to 36 weeks
  Treatment entry is determined by review of electronic medical record of whether clients attended their first scheduled treatment session
Number of treatment sessions attended during the three-month outpatient treatment program based on electronic medical record review | up to 36 weeks
  Number of treatment sessions that clients attend is determined by review of electronic medical record and calculating number of treatment sessions attended.
Number of participants who completed the three-month outpatient treatment program based on electronic medical record review | up to 36 weeks
  Completion of the three-month outpatient treatment program is determined by review of electronic medical record

SECONDARY OUTCOMES:
Change from baseline in client readiness to enter treatment on the University of Rhode Island Change Assessment Scale (URICA) at 1 hour post-intake | baseline and 1 hour post-intake
  The URICA is a validated, self-report measure of client readiness for treatment engagement. Possible scores range from 32 to 160 with higher scores indicative greater readiness to enter treatment. Change = (Hour 1 score - Baseline Score).
Score on therapeutic alliance on the Working Alliance Inventory (WAI) at 1-hour post-intake | 1 hour post-intake
  The WAI is a validated, self-report measure of client perceptions of the therapeutic process by assessing three sub scales: Goals, Bond, and Tasks. Possible scores on sub scales range from 12 to 84 with higher scores indicative of better therapeutic alliance.

OTHER OUTCOMES:
Change from baseline in organizational readiness to change on the Texas Christian University-Organizational Readiness to Change (TCU-ORC) at 1 year | baseline and 1 year
  The TCU-ORC is a validated, self-report measure of personnel perceptions of their organization's readiness and willingness to make changes. Possible scores range from 125 to 625 with higher scores indicative of more readiness to change. Change = (Year 1 score - Baseline Score).
Change from baseline in organizational readiness to change on the Readiness for Organizational Change (ROC) at 1 year | baseline and 1 year
  The ROC is a validated, self-report measure of personnel perceptions of their organization's readiness to change. Possible scores range from 25 to 155 with higher scores indicative of more readiness to change. Change = (Year 1 score - Baseline Score).
Change from baseline in organizational capability to change on the Change Process Capability Questionnaire (CPCQ) at Year 1 | baseline and 1 year
  The CPCQ is a validated, self-report measure of personnel perceptions of of their organization's capability to change. Possible scores range from 1 to 132 with higher scores indicative of more capability to make changes in the organization. Change = (Year 1 score - Baseline Score).

CONTACTS AND LOCATIONS:
Overall Officials: Margo Hurlocker, PhD, Principal Investigator — University of New Mexico
Locations (1):
- Turning Point Recovery Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results reported in a peer-reviewed publication, after deidentification (text, tables, figures, and appendices). Session audio recordings will not be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available starting in January 2025
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data. A data use agreement will be required, signed by the requesting investigator and their Authorized Organization Representation (AOR)/Signing Official (SO)

REFERENCES:
- [Derived] Hurlocker MC, Moyers TB, Hatch M, Curran G, McCrady B, Venner KL, Witkiewitz K. Effectiveness and feasibility of a motivational interviewing intake (MII) intervention for increasing client engagement in outpatient addiction treatment: an effectiveness-implementation hybrid design protocol. Addict Sci Clin Pract. 2023 Oct 21;18(1):63. doi: 10.1186/s13722-023-00412-y. PMID 37865777